CLINICAL TRIAL: NCT03376724
Title: Effectiveness of the Functional Exercises in Young Adults Chronic Low Back Pain: a Randomized Controlled Trial
Brief Title: Functional Exercises for Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Emilia Moreira, PT, Pfysiotherapist, MsC, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP 1.346.703
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional exercise (Experimental)
  Interventions: Other: Functional Exercise Protocol; Other: Minimal
- Control Group (Active Comparator)
  Interventions: Other: Minimal

INTERVENTIONS:
Other: Functional Exercise Protocol — Functional exercise protocol. This protocol started with corporal conscience exercise, breathing, abdominal activation, activities such as sitting, getting up, climbing stairs, reaching with arms, moving forward, bodyweight exercises, bridges and boards. This protocol will be performed during 12 weeks, two sessions per week.
  Arms: Functional exercise
Other: Minimal — Analgesic use when necessary and a single back scholl class

SUMMARY:
Non-specific low back pain is a common condition. Exercise is effective treatment for chronic low back pain. We hypothesized the functional exercise group will present pain reduction and functional improvement.

The purpose of this study is investigated the effectiveness of an functional exercise program for people with nonspecific chronic low back pain. Patients will be randomly divided into 2 groups: control group (minimal intervention - mini back school and analgesic) and group will receive a functional exercise protocol associated with minimal intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 50 years
* Low back pain for more than 3 months
* Low back pain with numeric pain scale between 3 - 8 cm
* Understand Portuguese well enough to be able to fill in the questionnaires

Exclusion Criteria:

* Inflammatory/rheumatological diseases, tumor, infection or vertebral fracture;
* Main pain as leg pain (eg: nerve root compression or herniated disc with radicular pain / radiculopathy, lateral and central stenosis)
* Less than 6 months after lumbar spine, lower limb or abdomen surgery
* Previous spinal surgery;
* Previous spinal infiltration for pain relief in the last 3 months;
* Several scoliosis;
* Litigation;
* Pregnancy;
* Fibromyalgia;
* People who had changed physical activity or undergone physical therapy in the previous 3 months;
* Presence of any contraindication to exercise;
* Planned travel in the next 12 weeks;
* Geographic inaccessibility.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-05-10 (Estimated); Study Completion 2018-11-10 (Estimated)

PRIMARY OUTCOMES:
Low back of pain intensity measured with Numeric Pain Rating Scale | Baseline, 6, 12 and 24 weeks
  It will be measured by the Brazilian version of the Numeric Pain Rating Scale (NPRS) 11 points. The NPRS goes from 0 to 10, where 0 is "no pain" and 10 is "the worst pain imaginable." Participants will be asked to answer about their pain levels based on the last seven days. Change in pain score or an improvement of 2 levels or more is accepted as clinically relevant.

SECONDARY OUTCOMES:
Disability associated to low back pain measured with Oswestry Disability Index | Baseline, 6, 12 and 24 weeks
  Change in Oswestry Disability Index score
Disability associated to low back pain measured with Roland Morris Disability | Baseline, 6, 12 and 24 weeks
  Change in Roland Morris Disability score
Fear of movement measured with Fear-Avoidance Beliefs Questionnaire | Baseline, 6, 12 and 24 weeks
  Change in Fear-Avoidance Beliefs Questionnaire score
Quality of life measured with Short form-36 questionnaire | Baseline, 6, 12 and 24 weeks
  Change in Short form-36 questionnaire score
Function measured with the 6-minute walk test | Baseline, 6, 12 and 24 weeks
  Change in 6-minute walk test
Function measured with the timed to up and go test | Baseline, 6, 12 and 24 weeks
  Change in timed to up and go test
Patient's global impression of recovery measured with a likert scale | 6, 12 and 24 weeks after baseline
  It will be evaluated based on the global perceived effect by the Likert Scale Score. The Likert scale, used to evaluate the patient's global perceived effect with treatment. The patients answered the question 'After starting the treatment, how do you think your low back is?' with one of the following statements: much worse, a little worse, unchanged, a little better, much better.
Analgesic consumption | 6, 12 and 24 weeks after baseline
  Change in analgesic consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Emilia Moreira, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No